CLINICAL TRIAL: NCT04562155
Title: Randomized, Double-blind, Parallel Group, Phase 2b Dose-finding, Efficacy and Safety Study of 12-week Twice Daily Oral Administration of BAY 1817080 Compared to Placebo in the Treatment of Refractory and/or Unexplained Chronic Cough (RUCC)
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Three Different Doses of BAY1817080 Compared to Placebo in Patients With Chronic Cough
Acronym: PAGANINI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20393; 2019-004169-42 (EudraCT Number)
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Results first posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-07

CONDITIONS: Refractory and/or Unexplained Chronic Cough
Keywords: RUCC; Chronic cough; P2X3 receptor antagonist
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BAY1817080 dose A BID (Experimental): Each participant will be randomized to receive one of three oral doses of BAY 1817080 or placebo, administered twice daily over the course of 12 weeks.
  Interventions: Drug: BAY1817080
- BAY1817080 dose B BID (Experimental): Each participant will be randomized to receive one of three oral doses of BAY 1817080 or placebo, administered twice daily over the course of 12 weeks.
  Interventions: Drug: BAY1817080
- BAY1817080 dose C BID (Experimental): Each participant will be randomized to receive one of three oral doses of BAY 1817080 or placebo, administered twice daily over the course of 12 weeks.
  Interventions: Drug: BAY1817080
- Placebo (Placebo Comparator): Each participant will be randomized to receive one of three oral doses of BAY 1817080 or placebo, administered twice daily over the course of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1817080 — Study drug BAY1817080 will be administered orally as tablet.
  Arms: BAY1817080 dose A BID; BAY1817080 dose B BID; BAY1817080 dose C BID
Drug: Placebo — Matching Placebo for BAY1817080 will be administered orally as tablet.
  Arms: Placebo

SUMMARY:
Researchers in this study want to find the optimal therapeutic dose of drug BAY1817080 for patients with long-standing cough with or without clear causes (refractory and/or unexplained chronic cough, RUCC). Study drug BAY1817080 is a new drug under development for the treatment of long-standing cough. It blocks proteins that are expressed by the airway sensory nerves which are oversensitive in patients with long-standing cough. This prevents the urge to cough. Researchers also want to learn the safety of the study drug and how well it works in reducing the cough frequency, severity and urge-to-cough.

Participants in this study will receive either the study drug or placebo (a placebo looks like the test drug but does not have any medicine in it) tablets twice daily for 12 weeks. Observation for each participant will last about 18 weeks in total. Participants will be asked to wear a digital device to record the cough and to complete questionnaires every day to document the symptoms. Blood samples will be collected from the participants to monitor the safety and measure the blood level of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age at the time of signing the informed consent.
* A cough that has lasted for at least 12 months (unresponsive to treatment options) with a diagnosis of refractory chronic cough and/or idiopathic (unexplained) chronic cough.
* Persistent cough for at least the last 8 weeks before screening.
* Women of childbearing potential must agree to use acceptable effective or highly effective birth control methods during the study and for at least 30 days after the last dose.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Smoking history within the last 12 months before screening (all forms of smoking, including e-cigarettes, cannabis and others), and any former smoker with more than 20 pack-years.
* Ongoing or previous exposure to inhalational toxic fumes (e.g., ammonia, chlorine, nitrogen dioxide, phosgene and sulfur dioxide) within the last 12 months before screening.
* Respiratory tract infection within 4 weeks before screening.
* History of chronic bronchitis.
* Systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg at screening visit.
* Positive SARS-CoV-2 virus RNA and/or serology IgG tests at screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (99):
- United States (8):
  - California Allergy & Asthma Medical Group & Research Center, Los Angeles, California
  - Florida Pediatrics, Largo, Florida
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - Minnesota Lung Center, Edina, Minnesota
  - Montana Medical Research, Inc, Missoula, Montana
  - Vanderbilt University Medical School, Nashville, Tennessee
  - Pharmaceutical Research & Consulting, Inc., Dallas, Texas
  - Bellingham Asthma, Allergy & Immunology Clinic, Bellingham, Washington
- Argentina (7):
  - Instituto Ave Pulmo, Mar del Plata, Buenos Aires
  - Centro Respiratorio Quilmes, Quilmes, Buenos Aires
  - Centro Médico Dra. De Salvo - Clinical Research Center, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Centro de Investigaciones Clínicas, CABA, Ciudad Auton. de Buenos Aires
  - Fundación CIDEA, CABA, Ciudad Auton. de Buenos Aires
  - Investigación en Alergias y Enfermedades Respiratorias-INAER, CABA, Ciudad Auton. de Buenos Aires
  - Investigaciones en Patologías Respiratorias, San Miguel de Tucumán, Tucumán Province
- Australia (5):
  - Macquarie University Hospital, Macquarie University, New South Wales
  - Maroubra Medical Centre, Maroubra, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Western Respiratory Trial Specialists, Spearwood, Western Australia
- Belgium (5):
  - Dr. MARTINOT Jean-Benoît, Erpent
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège, Liège
  - VZW Emmaus, Mechelen
- Canada (2):
  - Burlington Lung Clinic (BLC) Clinical Research, Burlington, Ontario
  - Clinique de pneumologie et du sommeil de Lanaudière (CPSL), Saint-Charles-Borromée, Quebec
- Czechia (5):
  - MUDr Otakar Hokynar - Plicni ambulance, Kralupy nad Vltavou
  - Ordinace pro TBC a respiracni nemoci, s.r.o., Olomouc
  - Dawon s.r.o., Prague
  - Plicní stredisko Teplice, s.r.o., Teplice
  - MUDr. Milan Sklenar, Varnsdorf
- France (2):
  - Cochin - Paris, Paris
  - CHU de Toulouse - Hôpital Larrey, Toulouse
- Germany (7):
  - Klinikum Konstanz, Konstanz, Baden-Wurttemberg
  - Zentrum f. ambulante pneumologische Forschung Marburg GbR, Marburg, Hesse
  - Ballenberger, Freytag, Wenisch, Neu-Isenburg, Hesse
  - Pneumologicum im Südstadt Forum, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Priv.-Doz. Dr. med. Christian Gessner, Leipzig, Saxony
  - Praxis f. Lungen- und Bronchialheilkunde,, Berlin
- Hungary (5):
  - D.Kenessey A Hospital, Balassagyarmat
  - EKBC, Uj Szent Janos Korhaz es Szakrendelo, Budapest
  - Erzsebet Gondozohaz, Gödöllő
  - Da Vinci Maganklinika, Pécs
  - Farmakontroll Bt., Százhalombatta
- Italy (4):
  - ASST Lodi, Lodi, Lombardy
  - A.O.U. Careggi, Florence, Tuscany
  - IRCCS Ospedale Sacro Cuore Don Calabria, Verona, Veneto
  - A.O.U.I. Verona, Verona, Veneto
- Japan (12):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - University of Fukui Hospital, Yoshida, Fukui
  - University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Idaimae Minami Yojo, Sapporo, Hokkaido
  - Japan community health care organization Kanazawa Hospital, Kanazawa, Ishikawa-ken
  - Komatsu Municipal Hospital, Komatsu, Ishikawa-ken
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital, Yokohama, Kanagawa
  - Matsusaka Municipal Hospital, Matsusaka, Mie-ken
  - Hamamatsu Rosai Hospital, Hamamatsu, Shizuoka
  - Tokyo Shinagawa Hospital, Shinagawa-ku, Tokyo
  - Fukushima Medical University Hospital, Fukushima
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Isala, Zwolle
- Poland (5):
  - Centrum Medycyny Oddechowej Mroz Spolka Jawna, Bialystok
  - KLIMED Marek Klimkiewicz, Bychawa
  - Centrum Alergologii Sp. z o.o., Lublin
  - Ostrowieckie Centrum Medyczne Sp. Cyw. A.O-C. K.C., Ostrowiec Świętokrzyski
  - Centrum Medyczne Lucyna Andrzej Dymek, Strzelce Opolskie
- Russia (7):
  - Region Clinical Emergency Hospital n.a. M.A.Podgorbunskogo, Kemerovo
  - City Clinical Hospital n.a. D.D. Pletnev, Moscow
  - LLC "Medical Center "SibNovoMed"", Novosibirsk
  - City Consultative and Diagnostic Center #1, Saint Petersburg
  - LLC Astarta, Saint Petersburg
  - City Clinical Hospital #4 Samara, Samara
  - Voronezh Regional Clinical Hospital #1, Voronezh
- Slovakia (5):
  - ALIAN s.r.o., Bardejov
  - INSPIRO, s.r.o., Humenné
  - AlergoImunocentrum, s.r.o., Kežmarok
  - Plucna ambulancia s.r.o., Poprad
  - Ambulancia klin. imunologie a alergologie, ANA JJ, s.r.o., Topoľčany
- Spain (3):
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
- Taiwan (5):
  - Chang Gung Memorial Hospital Keelung, Keelung
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
- Turkey (Türkiye) (5):
  - Akdeniz Universitesi Tip Fakultesi Hastanesi, Antalya
  - Istanbul Universitesi Cerrahpasa-Cerrahpasa Tip Fakultesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Sureyyapasa Gogus Hasalikleri. ve Gogus Cerrahisi EAH, Maltepe
  - Mersin Universitesi Tip Fakultesi, Mersin
- United Kingdom (5):
  - North Tyneside General Hospital, North Shields, Tyne and Wear
  - West Walk Surgery, Bristol
  - Castle Hill Hospital, Cottingham
  - King's College Hospital - NHS Foundation Trust, London
  - University Hospital of South Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Background] Fletcher MC. Selectivity of the P2X3 receptor antagonist Eliapixant, and its potential use in the treatment of endometriosis. Purinergic Signal. 2022 Mar;18(1):1-3. doi: 10.1007/s11302-021-09831-5. Epub 2022 Jan 3. No abstract available. PMID 34978027
- [Derived] Trigg A, Clarke N, Gerlinger C, Krahn U, Gater A, Haberland C. Psychometric validation of the severity of chronic cough diary, leicester cough questionnaire, and a cough severity visual analogue scale in patients with refractory chronic cough. J Patient Rep Outcomes. 2025 Jun 11;9(1):65. doi: 10.1186/s41687-025-00888-z. PMID 40498172
- [Derived] Dicpinigaitis PV, Morice AH, Smith JA, Sher MR, Vaezi M, Guilleminault L, Niimi A, Gude K, Krahn U, Saarinen R, Pires PV, Wosnitza M, McGarvey L; PAGANINI Investigators. Efficacy and Safety of Eliapixant in Refractory Chronic Cough: The Randomized, Placebo-Controlled Phase 2b PAGANINI Study. Lung. 2023 Jun;201(3):255-266. doi: 10.1007/s00408-023-00621-x. Epub 2023 Jun 1. PMID 37261531
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 99 centers in 19 countries/regions with first participant first visit on 02-Oct-2020 and last participant last visit on 23-Jul-2021.
Pre-assignment Details: Overall, 399 participants were screened, 89 of whom were screening failures. The remaining 310 participatns were randomized to 4 treatment groups (75 to eliapixant 25 mg BID, 78 to eliapixant 75 mg BID, 80 to eliapixant 150 mg BID, and 77 to placebo).
Groups:
- Eliapixant 25 mg BID: Participants were randomized to receive 25 mg oral doses of eliapixant, administered twice daily over the course of 12 weeks.
- Eliapixant 75 mg BID: Participants were randomized to receive 75 mg oral doses of eliapixant, administered twice daily over the course of 12 weeks.
- Eliapixant 150 mg BID: Participants were randomized to receive 150 mg oral doses of eliapixant, administered twice daily over the course of 12 weeks.
- Placebo: Participants were randomized to receive placebo for eliapixant, administered twice daily over the course of 12 weeks.
Period: Overall Study
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Started | 75 | 78 | 80 | 77
Completed | 64 | 69 | 67 | 71
Not Completed | 11 | 9 | 13 | 6
Not completed — COVID-19 pandemic | 0 | 0 | 0 | 1
Not completed — Adverse Event | 7 | 3 | 8 | 1
Not completed — Withdrawal by Subject | 3 | 6 | 3 | 3
Not completed — Participant personal reason | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo | Total
Number analyzed (Participants) | 75 | 78 | 80 | 77 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] — Used full analysis set: All participants randomly assigned to study intervention.
  years | 61.81 (9.64) | 58.62 (12.7) | 58.98 (11.8) | 56.91 (12.4) | 59.06 (11.79)
Age, Customized [Number; unit: Participants] — Used full analysis set
  Participants
    Adults (18-64 years) | 45 | 50 | 49 | 49 | 193
    From 65-84 years | 30 | 28 | 31 | 28 | 117
Sex: Female, Male [Count of Participants; unit: Participants] — Used full analysis set
  Participants
    Female | 56 | 63 | 61 | 61 | 241
    Male | 19 | 15 | 19 | 16 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Used full analysis set
  Participants
    Hispanic or Latino | 1 | 4 | 3 | 2 | 10
    Not Hispanic or Latino | 74 | 74 | 77 | 75 | 300
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline 24-hour coughs per hour [Geometric Mean (Standard Deviation); unit: 24-hour cough count per hour] — Used per protocol set (PPS): All participants randomly assigned to study intervention who did not have validity findings affecting efficacy. Participants were analyzed according to the intervention they actually received. If a participant received different interventions during the study, he/she was excluded from the PPS.
  The main reasons for excluding the participants from the PPS were that there was no valid post-baseline measurement available due to an intercurrent event (15 participants, 4.8%) or that the participant had used prohibited concomitant medication (9 participants, 2.9%). Population: Used per protocol set (PPS)
  24-hour cough count per hour
    number analyzed (Participants) | 67 | 69 | 73 | 74 | 283
    (all) | 17.49 (2.94) | 19.23 (2.94) | 15.61 (2.34) | 17.63 (3.07) | 17.42 (2.81)
Baseline Leicester Cough Questionnaire (LCQ) Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The LCQ was a 19-item instrument that asked about the impact of chronic cough on various aspects of participants' lives. 8 items built the physical domain. 7 items built the psychological domain. 4 items built the social domain. Study participants responded to the items using a 7-point Likert scale from 1 (all of the time) to 7 (none of the time) and entered their assessments on a tablet device. The LCQ total score was calculated as a mean score for each of the three domains ranging from 1 to 7, with the LCQ total score ranging from 3 to 21. Population: Used per protocol set (PPS)
  Scores on a scale
    number analyzed (Participants) | 67 | 69 | 73 | 74 | 283
    (all) | 12.00 (2.54) | 11.76 (2.77) | 11.15 (2.56) | 11.53 (3.27) | 11.60 (2.81)
Baseline awake cough count per hour [Geometric Mean (Standard Deviation); unit: Cough count per hour] — Population: Used per protocol set (PPS)
  Cough count per hour
    number analyzed (Participants) | 67 | 69 | 73 | 74 | 283
    (all) | 23.62 (3.02) | 26.41 (2.97) | 21.19 (2.39) | 24.01 (3.18) | 23.70 (2.88)
Baseline Cough Severity Visual Analogue Scale [VAS] Value [Mean (Standard Deviation); unit: Scores on a scale] — The Cough Severity VAS was a single item instrument, asking the study participant to assess the severity of his/her cough using a 0-100 VAS.
  This was a vertically oriented line ordered from 0-100, with 0 = "No Cough" and 100 = "Extremely Severe Cough". Population: Used per protocol set (PPS) - Included the participants in PPS with valid VAS value.
  Scores on a scale
    number analyzed (Participants) | 62 | 68 | 67 | 69 | 266
    (all) | 65.51 (14.64) | 67.08 (14.89) | 66.79 (15.86) | 61.52 (18.51) | 65.20 (16.16)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Cough Count After 12 Weeks of Intervention
Description: The raw 24-hour cough count measured by cough recording digital wearable monitoring device was standardized to an average hourly count. For the ratio between the geometric means of 24-hour cough count, the geometric mean of 24-hour cough count after 12 weeks of intervention was divided by the geometric mean of 24-hour cough count at baseline.
  btw = between geo = geometric
Time Frame: From baseline up to 12 weeks
Population: All participants in PPS with valid 24-hour cough count values in Week 12 or Termination visit.
Measure: Geometric Mean (Standard Deviation); unit: Ratio btw geoMeans of 24h cough count
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Number analyzed (Participants) | 64 | 68 | 72 | 73
Ratio btw geoMeans of 24h cough count | 0.56 (0.9191) [lower limit 0.9191] | 0.47 (0.9019) [lower limit 0.9019] | 0.52 (0.8608) [lower limit 0.8608] | 0.64 (0.7855) [lower limit 0.7855]
Statistical Analysis 1: Comparison: Eliapixant 25 mg BID vs Eliapixant 75 mg BID vs Eliapixant 150 mg BID vs Placebo; Detection of dose-response: Emax model (ED50=30) Dose response relationship was assessed using the MCP-Mod method combining multiple comparison procedures (MCP) principles with modeling techniques. A generalized MCP approach (with adjustment for baseline cough count and geographic region) was applied to calculate the adjusted one-sided p-values of the contrast test. Pre-specified overall Type one error at alpha level of 0.1 (one-sided); Test type: Superiority; p = 0.0345, MCP-Mod method — Adjusted p-value
Statistical Analysis 2: Comparison: Eliapixant 25 mg BID vs Eliapixant 75 mg BID vs Eliapixant 150 mg BID vs Placebo; Detection of dose-response: Emax model (ED50=50) Dose response relationship was assessed using the MCP-Mod method combining multiple comparison procedures (MCP) principles with modeling techniques. A generalized MCP approach (with adjustment for baseline cough count and geographic region) was applied to calculate the adjusted one-sided p-values of the contrast test. Pre-specified overall Type one error at alpha level of 0.1 (one-sided); Test type: Superiority; p = 0.0376, MCP-Mod method — Adjusted p-value
Statistical Analysis 3: Comparison: Eliapixant 25 mg BID vs Eliapixant 75 mg BID vs Eliapixant 150 mg BID vs Placebo; Detection of dose-response: sigm. Emax model (ED50=30, h=3) sigm = sigmoidal h = hill parameter Dose response relationship was assessed using the MCP-Mod method combining multiple comparison procedures (MCP) principles with modeling techniques. A generalized MCP approach (with adjustment for baseline cough count and geographic region) was applied to calculate the adjusted one-sided p-values of the contrast test. Pre-specified overall Type one error at alpha level of 0.1 (one-sided); Test type: Superiority; p = 0.0319, MCP-Mod method — Adjusted p-value
Statistical Analysis 4: Comparison: Eliapixant 25 mg BID vs Eliapixant 75 mg BID vs Eliapixant 150 mg BID vs Placebo; Detection of dose-response: sigm. Emax model (ED50=60, h=5) sigm = sigmoidal h = hill parameter Dose response relationship was assessed using the MCP-Mod method combining multiple comparison procedures (MCP) principles with modeling techniques. A generalized MCP approach (with adjustment for baseline cough count and geographic region) was applied to calculate the adjusted one-sided p-values of the contrast test. Pre-specified overall Type one error at alpha level of 0.1 (one-sided); Test type: Superiority; p = 0.0603, MCP-Mod method — Adjusted p-value

2. Secondary Outcome: Percentage of Participants With a ≥30% Reduction From Baseline in 24-hour Cough Count After 12 Weeks of Intervention
Description: The raw 24-hour cough count measured by cough recording digital wearable monitoring device was standardized to an average hourly count. The change from baseline in 24-hour cough count was calculated by the geometric mean of 24-hour cough count after 12 weeks of intervention minus the geometric mean at baseline divided by the geometric mean at baseline. The percentage of participants with a reduction of ≥30% is shown
Time Frame: From baseline up to 12 weeks
Population: PPS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 73 | 74
Percentage of participants | 52.24 (39.67) [39.67 to 64.60] | 63.77 (51.31) [51.31 to 75.01] | 53.42 (41.37) [41.37 to 65.20] | 45.95 (34.29) [34.29 to 57.93]

3. Secondary Outcome: Change From Baseline in 24-hour Cough Count After 2, 4, and 8 Weeks of Intervention
Description: The raw 24-hour cough count measured by cough recording digital wearable monitoring device was standardized to an average hourly count. For the ratio between the geometric means of 24-hour cough count, the geometric mean of 24-hour cough count after 2, 4, and 8 weeks of intervention was divided by the geometric mean of 24-hour cough count at baseline.
  btw = between geo = geometric
Time Frame: From baseline up to 2 weeks, 4 weeks and 8 weeks
Population: PPS
Measure: Geometric Mean (Standard Deviation); unit: Ratio btw geoMeans of 24h cough count
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 73 | 74
Ratio btw geoMeans of 24h cough count
  Week 2: number analyzed (Participants) | 65 | 67 | 72 | 73
  Week 2 | 0.75 (0.6134) | 0.58 (0.8209) | 0.61 (0.6636) | 0.75 (0.4762)
  Week 4: number analyzed (Participants) | 66 | 66 | 68 | 71
  Week 4 | 0.64 (0.7237) | 0.51 (0.8192) | 0.58 (0.8589) | 0.69 (0.6657)
  Week 8: number analyzed (Participants) | 64 | 65 | 69 | 72
  Week 8 | 0.55 (0.8737) | 0.46 (0.9484) | 0.51 (0.8827) | 0.70 (0.6451)

4. Secondary Outcome: Change From Baseline in Awake Cough Frequency Per Hour After 2, 4, 8 and 12 Weeks of Intervention
Description: Measured by cough recording digital wearable monitoring device
  btw = between geo = geometric
Time Frame: From baseline up to 2 weeks, 4 weeks, 8 weeks and 12 weeks
Population: PPS
Measure: Geometric Mean (Standard Deviation); unit: Ratio btw geoMeans of 24h cough count
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 73 | 74
Ratio btw geoMeans of 24h cough count
  Week 2: number analyzed (Participants) | 65 | 67 | 72 | 73
  Week 2 | 0.78 (0.6324) | 0.60 (0.8295) | 0.60 (0.6695) | 0.77 (0.4660)
  Week 4: number analyzed (Participants) | 66 | 66 | 68 | 71
  Week 4 | 0.67 (0.7390) | 0.53 (0.8128) | 0.57 (0.8983) | 0.72 (0.6637)
  Week 8: number analyzed (Participants) | 64 | 65 | 69 | 72
  Week 8 | 0.55 (0.9274) | 0.47 (0.9576) | 0.50 (0.9154) | 0.72 (0.6698)
  Week 12: number analyzed (Participants) | 64 | 68 | 72 | 73
  Week 12 | 0.56 (0.9582) | 0.47 (0.9051) | 0.47 (1.1338) | 0.65 (0.7926)

5. Secondary Outcome: Change From Baseline in Cough Related Quality of Life After 12 Weeks of Intervention
Description: Measured by Leicester Cough Questionnaire (LCQ) total score. The LCQ was a 19-item instrument that asked about the impact of chronic cough on various aspects of participants' lives using a recall period of two weeks. The 8 items: 1, 2, 3, 9, 10, 11, 14, 15 built the physical domain. 7 items: 4, 5, 6, 12, 13, 16, 17 built the psychological domain. Further 4 items: 7, 8, 18 and 19 built the social domain. Study participants responded to the items using a 7-point Likert scale from 1 (all of the time) to 7 (none of the time) and entered their assessments on a tablet device. Completion of the LCQ took approximately five minutes. The LCQ total score was calculated as a mean score for each of the three domains ranging from 1 to 7, with the LCQ total score ranging from 3 to 21.
Time Frame: From baseline up to 12 weeks
Population: All participants in PPS with valid Leicester Cough Questionnaire scores in Week 12 or Termination visit were included.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 72 | 74
Scores on a scale | 2.18 (3.44) [lower limit 3.44] | 2.50 (3.29) [lower limit 3.29] | 2.73 (3.53) [lower limit 3.53] | 2.16 (3.12) [lower limit 3.12]

6. Secondary Outcome: Change From Baseline in Cough Severity After 12 Weeks of Intervention
Description: Measured by Cough Severity Visual Analogue Scale (VAS). The Cough Severity VAS was a single item instrument, asking the study participant to assess the severity of his/her cough using a 0-100 VAS.
  This was a vertically oriented line ordered from 0-100, with 0 = "No Cough" and 100 = "Extremely Severe Cough".
Time Frame: From baseline up to 12 weeks
Population: All participants in PPS with valid VAS scores in Week 12 or Termination visit.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Number analyzed (Participants) | 61 | 68 | 67 | 68
Scores on a scale | -17.69 (23.87) [lower limit 23.87] | -22.66 (22.98) [lower limit 22.98] | -22.87 (24.54) [lower limit 24.54] | -17.02 (21.88) [lower limit 21.88]

7. Secondary Outcome: Percentage of Participants With a ≥30 Scale Units Reduction From Baseline After 12 Weeks of Intervention
Description: Measured by cough Severity VAS
Time Frame: From baseline up to 12 weeks
Population: PPS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 73 | 74
Percentage of participants | 26.87 (16.76) [16.76 to 39.10] | 36.23 (24.99) [24.99 to 48.69] | 27.40 (17.61) [17.61 to 39.09] | 20.27 (11.81) [11.81 to 31.22]

8. Secondary Outcome: Percentage of Participants With a ≥1.3-point Increase From Baseline After 12 Weeks of Intervention
Description: Measured by LCQ total score. The LCQ was a 19-item instrument that asked about the impact of chronic cough on various aspects of participants' lives using a recall period of two weeks. The 8 items: 1, 2, 3, 9, 10, 11, 14, 15 built the physical domain. 7 items: 4, 5, 6, 12, 13, 16, 17 built the psychological domain. Further 4 items: 7, 8, 18 and 19 built the social domain. Study participants responded to the items using a 7-point Likert scale from 1 (all of the time) to 7 (none of the time) and entered their assessments on a tablet device. Completion of the LCQ took approximately five minutes. The LCQ total score was calculated as a mean score for each of the three domains ranging from 1 to 7, with the LCQ total score ranging from 3 to 21. The percentage of participants with a >= 1.3-point increase in LCQ total score is shown.
Time Frame: From baseline up to 12 weeks
Population: PPS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Number analyzed (Participants) | 67 | 69 | 73 | 74
Percentage of participants | 47.76 (35.40) [35.40 to 60.33] | 60.87 (48.37) [48.37 to 72.40] | 64.38 (52.31) [52.31 to 75.25] | 51.35 (39.44) [39.44 to 63.15]

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Associated Severity
Description: Adverse event (AE) was defined as any untoward medical occurrence in a study participant, whether or not considered related to the study intervention, occurring from the time of signing the informed consent until the follow-up visit.
  TEAE was defined as any event occurring or worsening after the start of study intervention administration until 14 days after the last intake of study intervention.
Time Frame: From the start of study intervention administration until 14 days after the last study medication intake, with an average of 80.0 + 14 days
Population: Safety analysis set (SAF): All participants randomly assigned to study intervention and who took at least one tablet of study intervention. Participants were analyzed according to the intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
Number analyzed (Participants) | 75 | 78 | 80 | 77
Participants
  Any TEAE | 43 | 51 | 51 | 39
  Maximum intensity for any TEAE - mild | 21 | 32 | 23 | 18
  Maximum intensity for any TEAE - moderate | 22 | 16 | 25 | 20
  Maximum intensity for any TEAE - severe | 0 | 3 | 3 | 1
  Any serious TEAE | 0 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: From the start of study intervention administration until 14 days after the last study medication intake, with an average of 80.0 + 14 days. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, with an average of 80.0 + 30 ± 5 days.
Arm/Group | Eliapixant 25 mg BID | Eliapixant 75 mg BID | Eliapixant 150 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/78 | 0/80 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/78 | 2/80 | 1/77
Other Adverse Events (participants affected / at risk) | 32/75 | 37/78 | 45/80 | 25/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eliapixant 25 mg BID (N=75) | Eliapixant 75 mg BID (N=78) | Eliapixant 150 mg BID (N=80) | Placebo (N=77)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eliapixant 25 mg BID (N=75) | Eliapixant 75 mg BID (N=78) | Eliapixant 150 mg BID (N=80) | Placebo (N=77)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 4 (5)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 5 (5) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 6 (6) | 5 (6) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood fibrinogen increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 9 (9) | 13 (14) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 5 (10) | 6 (7) | 4 (4)
Hypogeusia (Nervous system disorders) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7) | 7 (7) | 3 (3)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT04562155/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04562155/SAP_001.pdf